CLINICAL TRIAL: NCT03132480
Title: Study on TFA-1 Adhesive Forehead Sensors to Predict Fluid Responsiveness in Pediatric Patients Undergoing General Anesthesia
Brief Title: Fluid Responsiveness Using Forehead Sensor in Children
Acronym: forehead
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: H1703-137-841
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hypovolemia (Experimental)
  Interventions: Other: fluid resuscitation

INTERVENTIONS:
Other: fluid resuscitation — when the patients showed the clinical signs of hypovolemia, the fluid resuscitation with 10ml/kg crystalloid solution was performed.

SUMMARY:
Forehead sensor can predict the more accurate fluid responsiveness than finger sensor in children

DETAILED DESCRIPTION:
The investigator hypothesized that the forehead sensor can predict the fluid responsiveness more accurate than the finger sensor in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia for neurosurgery, major abdominal surgery, and cardiac surgical procedures.

Exclusion Criteria:

* preoperative Ejection fraction <30%
* underlying lung disease
* cardiac arrhythmia

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Area under the Receiver operating characteristic(ROC) curve (AUC) | before fluid resuscitation
  the predictability of fluid responsiveness was calculated using ROC analysis

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim EH, Kim H, Lee JH, Kim JT, Jang YE, Ji SH, Kim HS. Role of TFA-1 adhesive forehead sensors in predicting fluid responsiveness in anaesthetised children: A prospective cohort study. Eur J Anaesthesiol. 2020 Aug;37(8):713-718. doi: 10.1097/EJA.0000000000001235. PMID 32412989